CLINICAL TRIAL: NCT00003375
Title: A Phase II Study of Observation in Favorable Low-Grade Glioma and a Phase II Study of Radiation With or Without PCV Chemotherapy in Unfavorable Low-Grade Glioma
Brief Title: Observation or Radiation Therapy With or Without Combination Chemotherapy in Treating Patients With Low-Grade Glioma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); SWOG Cancer Research Network (Network); North Central Cancer Treatment Group (Network); Eastern Cooperative Oncology Group (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9802; CDR0000066367; E-R9802; NCCTG-R9802; SWOG-R9802
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult oligodendroglioma; adult diffuse astrocytoma; adult pilocytic astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma; Astrocytoma | interventions — Lomustine; Procarbazine; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Observation (No Intervention): Observation only.
- Radiation therapy (Experimental): Radiation therapy only.
  Interventions: Radiation: radiation therapy
- Radiation plus PCV chemotherapy (Experimental): Radiation and Procarbazine/CCNU/Vincristine (PCV) chemotherapy
  Interventions: Drug: lomustine; Drug: procarbazine hydrochloride; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Drug: lomustine
  Arms: Radiation plus PCV chemotherapy
Drug: procarbazine hydrochloride
  Arms: Radiation plus PCV chemotherapy
Drug: vincristine sulfate
  Arms: Radiation plus PCV chemotherapy
Radiation: radiation therapy
  Arms: Radiation plus PCV chemotherapy; Radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether radiation therapy combined with chemotherapy is more effective than radiation therapy alone in treating patients with low-grade glioma.

PURPOSE: Phase II/III trial to evaluate observation and to compare the effectiveness of radiation therapy with or without combination chemotherapy in treating patients with low-grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Identify the overall survival of low-risk adult patients with supratentorial low-grade glioma who are observed postoperatively.
* Compare the overall survival of high-risk adult patients with supratentorial low-grade glioma who receive postoperative external beam radiotherapy with or without procarbazine, lomustine, and vincristine (PCV) chemotherapy.
* Compare the toxic effects of postoperative radiotherapy with or without PCV chemotherapy in patients with unfavorable low-grade glioma.

OUTLINE: This is a randomized study. Patients are stratified according to tumor subtype (astrocytoma [mixed-astro dominant or equal astro/oligo mix] vs oligodendroglioma [mixed-oligo dominant]), age (younger than 40 vs at least 40), Karnofsky performance status (60-80% vs 90-100%), and contrast enhancement on preoperative scan (present vs absent). Patients with low-risk disease (younger than 40 years old whose tumors have been surgically removed) are assigned to arm I. Patients with high-risk disease (at least 40 years old or who have had incomplete tumor removal) are randomized to arm II or III.

* Arm I (low-risk patients): Patients are observed. Patients may receive treatment if tumor recurs.
* Arm II (high-risk patients): Patients receive daily external beam radiotherapy 5 days a week for 6 weeks.
* Arm III (high-risk patients): Patients receive radiotherapy as in arm II followed by chemotherapy 1 month later. Chemotherapy consists of oral lomustine on day 1, vincristine IV on days 8 and 29, and oral procarbazine on days 8-21. Each course of chemotherapy lasts 8 weeks. Patients may receive up to 6 courses of chemotherapy.

Patients are followed every 4 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 252 patients will be accrued within 5.25 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unifocal or multifocal supratentorial WHO grade II astrocytoma (diffuse fibrillary, protoplasmic, or gemistocytic), oligodendroglioma, or oligoastrocytoma
* Patients with neurofibromatosis are eligible
* No other low-grade histologies, including:

  * Pilocytic astrocytoma
  * Subependymal giant cell astrocytoma of tuberous sclerosis
  * Subependymoma
  * Pleomorphic xanthoastrocytoma
  * Presence of a neuronal element such as ganglioglioma
  * Dysneuroembryoplastic epithelial tumor
* No presence of any high-grade glioma, including:

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Anaplastic oligodendroglioma
  * Anaplastic oligoastrocytoma
* No tumors in nonsupratentorial or other locations including optic chiasm, optic nerve(s), pons, medulla, cerebellum, or spinal cord
* No evidence of spread to spinal meninges or noncontiguous cranial meninges (i.e., leptomeningeal gliomatosis)
* No gliomatosis cerebri

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Hematopoietic:

* For high-risk patients:

  * Granulocyte count at least 1,500/mm^3
  * Platelet count normal

Hepatic:

* Bilirubin no greater than 2 times normal
* SGOT or SGPT no greater than 4 times normal
* Alkaline phosphatase no greater than 2 times normal

Renal:

* Creatinine no greater than 2 times normal

Pulmonary:

* No chronic lung disease (unless DLCO at least 60%)

Neurological:

* Neurologic function score no greater than 3

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or nonmelanoma skin cancer
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* No prior radiotherapy to the head or neck (unless brain is clearly excluded, such as radiotherapy for localized vocal cord cancer)

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 1998-10; Primary Completion 2005-08 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Overall Survival | From randomization to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 5 years or 80 deaths have been reported.

SECONDARY OUTCOMES:
Progression-free Survival | From randomization to the date of progression, death or last follow-up. Analysis ours at the same time as the primary outcome analysis.
The severe or worse toxicities (>= grade 3) of unfavorable patients | From start of treatment to end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Edward G. Shaw, MD, Study Chair — Wake Forest University Health Sciences; Geoffrey R. Barger, MD, Study Chair — Barbara Ann Karmanos Cancer Institute; Jan C. Buckner, MD, Study Chair — Mayo Clinic; Minesh P. Mehta, MD, Study Chair — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: Yes
Individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

REFERENCES:
- [Result] Prabhu RS, Won M, Shaw EG, Hu C, Brachman DG, Buckner JC, Stelzer KJ, Barger GR, Brown PD, Gilbert MR, Mehta MP. Effect of the addition of chemotherapy to radiotherapy on cognitive function in patients with low-grade glioma: secondary analysis of RTOG 98-02. J Clin Oncol. 2014 Feb 20;32(6):535-41. doi: 10.1200/JCO.2013.53.1830. Epub 2014 Jan 13. PMID 24419119
- [Result] Shaw EG, Wang M, Coons SW, Brachman DG, Buckner JC, Stelzer KJ, Barger GR, Brown PD, Gilbert MR, Mehta MP. Randomized trial of radiation therapy plus procarbazine, lomustine, and vincristine chemotherapy for supratentorial adult low-grade glioma: initial results of RTOG 9802. J Clin Oncol. 2012 Sep 1;30(25):3065-70. doi: 10.1200/JCO.2011.35.8598. Epub 2012 Jul 30. PMID 22851558
- [Result] Shaw EG, Berkey B, Coons SW, Bullard D, Brachman D, Buckner JC, Stelzer KJ, Barger GR, Brown PD, Gilbert MR, Mehta M. Recurrence following neurosurgeon-determined gross-total resection of adult supratentorial low-grade glioma: results of a prospective clinical trial. J Neurosurg. 2008 Nov;109(5):835-41. doi: 10.3171/JNS/2008/109/11/0835. PMID 18976072
- [Result] Shaw EG, Wang S, Coons S, et al.: Final report of Radiation Therapy Oncology Group (RTOG) protocol 9802: radiation therapy (RT) versus RT + procarbazine, CCNU, and vincristine (PCV) chemotherapy for adult low-grade glioma (LGG). [Abstract] J Clin Oncol 26 (Suppl 15): A-2006, 2008.
- [Result] Shaw EG, Berkey B, Coons SW, et al.: Initial report of Radiation Therapy Oncology Group (RTOG) 9802: prospective studies in adult low-grade glioma (LGG). [Abstract] J Clin Oncol 24 (Suppl 18): A-1500, 2006.
- [Derived] Bell EH, Zhang P, Shaw EG, Buckner JC, Barger GR, Bullard DE, Mehta MP, Gilbert MR, Brown PD, Stelzer KJ, McElroy JP, Fleming JL, Timmers CD, Becker AP, Salavaggione AL, Liu Z, Aldape K, Brachman DG, Gertler SZ, Murtha AD, Schultz CJ, Johnson D, Laack NN, Hunter GK, Crocker IR, Won M, Chakravarti A. Comprehensive Genomic Analysis in NRG Oncology/RTOG 9802: A Phase III Trial of Radiation Versus Radiation Plus Procarbazine, Lomustine (CCNU), and Vincristine in High-Risk Low-Grade Glioma. J Clin Oncol. 2020 Oct 10;38(29):3407-3417. doi: 10.1200/JCO.19.02983. Epub 2020 Jul 24. PMID 32706640
- [Derived] Buckner JC, Shaw EG, Pugh SL, Chakravarti A, Gilbert MR, Barger GR, Coons S, Ricci P, Bullard D, Brown PD, Stelzer K, Brachman D, Suh JH, Schultz CJ, Bahary JP, Fisher BJ, Kim H, Murtha AD, Bell EH, Won M, Mehta MP, Curran WJ Jr. Radiation plus Procarbazine, CCNU, and Vincristine in Low-Grade Glioma. N Engl J Med. 2016 Apr 7;374(14):1344-55. doi: 10.1056/NEJMoa1500925. PMID 27050206
- See also: Related Info — https://nctn-data-archive.nci.nih.gov/